CLINICAL TRIAL: NCT05865483
Title: A Multidimensional Profile of Dysphagia in People Living With Myotonic Dystrophy Type 1 (plwDM1)
Brief Title: Profile of Dysphagia in Myotonic Dystrophy Type 1 (DM1)
Acronym: SwallowDM1
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Myotonic Dystrophy Support Group, United Kingdom (Unknown); The National Brain Appeal, The National Hospital for Neurology and Neurosurgery (Unknown)
Responsible Party: Sponsor
Other Study IDs: 153848
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Myotonic Dystrophy 1; Dysphagia, Oropharyngeal
MeSH Terms: conditions — Myotonic Dystrophy; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Participant group: mild disease: Muscle impairment rating score (MIRS) (Mathieu et al., 2001) 1-2 (n=30)
- Participant group: moderate disease: Muscle impairment rating score (MIRS) (Mathieu et al., 2001) 3 (n=30)
- Participant group: severe disease: Muscle impairment rating score (MIRS) (Mathieu et al., 2001) 4-5 (n=30)
- Control group: No disease (n=60) age and sex-matched
- Caregiver group: Spends at least one mealtime daily assisting with a person with DM1 already enrolled in the study. Expect ratio of 1:2 caregiver:participant (approx n=45)

SUMMARY:
The goal of this observational study is to learn about swallowing difficulties (dysphagia) in patients living with myotonic dystrophy type 1 (DM1). The main questions it aims to answer are:

* whether the size and structure of the muscles involved in swallowing differ to those without the disease
* how the size and structure of muscles may associate with swallowing function and swallowing symptoms in this group.

Participants will undergo a range of tests including:

* Ultrasound (US) assessment of the muscles involved in swallowing
* An x-ray swallowing study (known as videofluoroscopy)
* Assessment of swallowing symptoms, including questionnaires
* Assessments of mobility, activity and breathing
* Assessments of quality of life and wellbeing

DETAILED DESCRIPTION:
This study will explore swallowing difficulties (dysphagia) caused by Myotonic Dystrophy Type 1 (DM1). Dysphagia causes food, drink and saliva to travel onto the lungs (aspiration) and can lead to pneumonia. Aspiration pneumonia is frequent and accounts for over 40% of deaths in DM1. Dysphagia also causes fear and anxiety which can lead to permanent lifestyle changes.

A better understanding of dysphagia in DM1 will improve our assessment and treatment and reduce its life-changing consequences. This research aims to define the dysphagia profile of people with DM1 (pwDM1) across the domains of structure, function, experience, and wellbeing by:

1. Investigating the size and structure of muscles involved in swallowing in patients with and without DM1.
2. Exploring how muscle size and structure are associated with i) swallowing function and ii) symptoms
3. Exploring how swallowing function is associated with i) symptoms, ii) patient and caregiver wellbeing and iii) other aspects of DM1 such as walking and breathing.

People aged 18+ with a confirmed diagnosis of DM1 will be invited to take part. Approximately 90 pwDM1 will be recruited. They will undergo a battery of tests including:

* Ultrasound (US) assessment of the muscles involved in swallowing
* An x-ray swallowing study (known as videofluoroscopy)
* Assessment of swallowing symptoms, including questionnaires
* Assessments of mobility, activity and breathing
* Assessments of quality of life and wellbeing

A sub-group of 20 pwDM1 will also undergo magnetic resonance imaging (MRI) of the muscles involved in swallowing to examine in detail the changes in seen on ultrasound. Approximately 60 people without DM1 will act as a control group for the US assessments. Primary caregivers of those with DM1 will be invited to complete a wellbeing questionnaire.

Data will be analysed using statistical methods and findings will be used to develop clinical practice recommendations for the assessment and treatment of dysphagia in DM1.

This study is part of an NIHR-funded clinical doctoral research fellowship (CDRF) and will take place at The National Hospital for Neurology and Neurosurgery (NHNN) in London. The maximum timescale for the study from opening recruitment to data collection of the final participant is 18 months (approx. 1st April 2023 - 30th September 2024).

ELIGIBILITY:
Participants with DM1

Inclusion:

* ≥18 years of age
* genetically confirmed of DM1
* able to eat & drink at least five sips of liquid by mouth at one time.

Exclusion:

* any condition or treatment other than DM1 that potentially influences swallowing muscle composition or function (e.g., a history of stroke or throat cancer).
* any patients who are pregnant
* patients with congenital or childhood DM1
* patients who are not able to eat or drink anything by mouth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with DM1, with and without reported swallowing difficulties, and relevant (age and sex-matched) controls. To ensure a spectrum of disease, participants will be recruited to one of three groups (mild, moderate, severe) according to the severity of their neuromuscular disability. Participants with DM1 must be taking food/drink by mouth (minimum five sips of fluid at a time).
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Swallowing muscle (geniohyoid) size | 16 months
Swallowing muscle (geniohyoid) structure | 16 months

SECONDARY OUTCOMES:
Association between muscle (size and structure) and dynamic swallowing assessment (VFSS) | 16 months
Association between muscle (size and structure) and strength (Iowa Oral Performance Instrument & bite-force) | 16 months
Association between muscle (size and structure) and swallowing speed (timed water swallow test & timed test of mastication) | 16 months
Association between muscle (size and structure) and patient symptoms (Sydney Swallow Questionnaire & SWAL-QOL) | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Taylor, PhD, Principal Investigator — University College London & University College London Hospitals
Locations (1):
- The National Hospital for Neurology & Neurosurgery, University College London Hospitals, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathieu J, Boivin H, Meunier D, Gaudreault M, Begin P. Assessment of a disease-specific muscular impairment rating scale in myotonic dystrophy. Neurology. 2001 Feb 13;56(3):336-40. doi: 10.1212/wnl.56.3.336. PMID 11171898